CLINICAL TRIAL: NCT05951816
Title: Phase 1 Study to Investigate the Dosimetry and Biodistribution of a Single Intravenous Administration of 99mTc-p5+14 Using SPECT/CT Imaging and Planar Gamma Scintigraphy in Healthy Volunteers and Patients With AL or ATTR Systemic Amyloidosis
Brief Title: A Phase 1 Study of 99mTc-p5+14 in Healthy Volunteers and Patients With AL or ATTR Systemic Amyloidosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Collaborators: Attralus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UTGSM-164388-101
Record Dates: First submitted 2023-06-30; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Systemic Amyloidosis
Keywords: Amyloidosis; p5+14; SPECT imaging; iodine-124-evuzamitide
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — Technetium; Technetium Tc 99m Pyrophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Estimation of dosimetry for 99mTc-p5+14 and Biodistribution Of 99mtc-p5+14 In Healthy Subjects (Experimental): For dosimetry, patients with a confirmed diagnosis of systemic AL amyloidosis, patients will be administered a single IV dose of up to 1 mg of 99mTc-p5+14 (~20 mCi) by slow push (~1 mL/5 sec.). Patients will then undergo serial planar scintigraphic imaging at ~30 minutes, ~1 hour, ~2 hours, ~4 hours, ~6 hours, and ~24 hours post-injection. At the 4-hour time point, the patient will also undergo a single SPECT/CT scan to provide additional data for estimating dosimetry. Before injection of the radiotracer and at each imaging session, ~2 -3 mL of blood will be acquired to determine the whole blood radioactivity.
  Healthy volunteers will undergo an echo examination, thereafter, they will be administered a single IV dose of 99mTc-p5+14 (20 mCi) and will undergo a single planar image acquisition followed by SPECT/CT imaging at ~1 hour and ~3 hours post-injection.
  Interventions: Drug: 99mTc-p5+14 is an amyloid reactive peptide labeled with technetium-99m.
- Biodistribution in patients with systemic AL or ATTR amlyoidosis (Experimental): Patients with a confirmed diagnosis of systemic AL or ATTR (with or without a positive PyP scan) will be administered a single IV dose of up to 1 mg of 99mTc-p5+14 (~20 mCi) by slow push (~1 mL/5 sec.). At ~1 hour and ~3 hours post-injection, patients will undergo abdominothoracic planar imaging followed by SPECT/CT imaging covering the same area. Vital signs (blood pressure, respiration rate, temperature, and pulse) will be acquired before injection of the 99mTc-p5+14, and at ~3 hours post injection.
  On Day 3, patient will undergo a trans thoracic echo examination. On Day 4, patients will undergo Technescan™ 99mTc-PYP (20 mCi) planar and SPECT/CT imaging at ~1 hour and ~3 hours post-injection. Vital signs (blood pressure, respiration rate, temperature, and pulse) will be acquired before injection of the 99mPYP, and at ~3 hours post injection.
  Interventions: Drug: 99mTc-Pyrophosphate and 99mtc-p5+14 - an Amyloid Reactive Peptide Labeled With Technetium-99m.

INTERVENTIONS:
Drug: 99mTc-p5+14 is an amyloid reactive peptide labeled with technetium-99m. — Peptide p5+14 is a pan-amyloid reactive, synthetic 45 L-amino acid polypeptide with a net +12 positive charge that can bind two major components of all extracellular amyloid deposits: (i) hypersulfated heparan sulfate glycosaminoglycans (proteoglycans) and (ii) amyloid fibrils. The polypeptide, labeled with iodine-124, has been shown (study AMY1001) to bind amyloid in all organs including the heart. This study will evaluate a Tc-99m-labeled version of the peptide for gamma imaging.
  Arms: Estimation of dosimetry for 99mTc-p5+14 and Biodistribution Of 99mtc-p5+14 In Healthy Subjects
Drug: 99mTc-Pyrophosphate and 99mtc-p5+14 - an Amyloid Reactive Peptide Labeled With Technetium-99m. — 99mTc-PYP is an FDA-approved, commercially available bone-seeking radiotracer used routinely in nuclear medicine. 99mTC-PYP imaging is used clinically for the diagnosis of cardiac ATTR amyloidosis.
  Other Names: 99mTc-PYP
  Arms: Biodistribution in patients with systemic AL or ATTR amlyoidosis

SUMMARY:
This study will investigate 99mTc-p5+14, an amyloid-reactive synthetic peptide, p5+14, radiolabeled with technetium-99m, as a radiotracer for detecting paamyloid deposits in patients with AL or ATTR-associated systemic amyloidosis, notably with cardiac involvement.

DETAILED DESCRIPTION:
The University of Tennessee Graduate School of Medicine (UTGSM) is investigating 99mTc-p5+14, an amyloid-reactive synthetic peptide, p5+14, radiolabeled with technetium-99m, as a radiotracer for planar gamma scintigraphy (PGS), single photon emission computed tomography (SPECT) or SPECT with x-ray computed tomography (SPECT/CT) for the diagnosis of systemic amyloidosis, notably with cardiac involvement. Based on nonclinical data and clinical data of 124I-p5+14 from Study AMY1001, peptide p5+14 binds many types of human amyloid and is rapidly cleared from the central compartment. When radiolabeled with 99mTc, p5+14 may enable visualization of amyloid laden tissues and organs by SPECT/CT imaging or PGS. Thus, this study has been designed to evaluate the dosimetry and biodistribution of 99mTc-p5+14 in patients with systemic amyloidosis compared with the biodistribution in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

PART 1

1. Understand the study procedures and agree to participate in the study by giving written informed consent as described in Section 10.1 - Appendix 1.
2. Be male or female >18 years of age.
3. Women of child-bearing potential (WOCBP) (those who have not been surgically sterilized, are not postmenopausal [i.e., last menstrual period >2 years ago without pharmaceutical intervention], and women who are fertile) must have a negative pregnancy test prior within 24 h prior to infusion.
4. WOCBP who are not exclusively in same-sex relationships and male participants with female sexual partners who are WOCBP must agree to use adequate contraceptive methods, defined as use of a condom by the male partner combined with use of a highly effective method of contraception by the female partner, for at least 2.5 days after injection of 99mTc-p5+14.
5. Have a confirmed diagnosis of systemic AL amyloidosis based on either a histologic confirmation with a biopsy containing deposits of apple-green birefringent, Congophilic material with aberrant organ-specific biomarkers indicating amyloid involvement, physical examination, or imaging study.
6. Have a diagnosis of cardiac amyloidosis within 2 years of screening. PART 2

1) Understand the study procedures and agree to participate in the study by giving written informed consent as described in Section 10.1 - Appendix 1.

2) Be male or female >18 years of age. 3) WOCBP (those who have not been surgically sterilized, are not postmenopausal [i.e., last menstrual period > 2 years ago without pharmaceutical intervention], and women who are fertile) must have a negative pregnancy test prior within 24 h prior to infusion.

4) WOCBP who are not exclusively in same-sex relationships and male participants with female sexual partners who are WOCBP must agree to use adequate contraceptive methods, defined as use of a condom by the male partner combined with use of a highly effective method of contraception by the female partner, for at least 2.5 days after injection of 99mTc-p5+14.

5) Have one of the following:

1. a confirmed diagnosis of systemic AL amyloidosis, based on either a histologic confirmation of a cardiac or extracardiac biopsy containing deposits of apple-green birefringent, Congophilic material AND imaging parameters (ECHO or CMR) indicative of cardiac involvement.
2. a confirmed diagnosis of systemic ATTR amyloidosis, based on either a histologic confirmation of a cardiac biopsy containing deposits of apple-green birefringent, Congophilic material or extracardiac biopsy and imaging parameters (ECHO or CMR or 99mTc-PYP) indicative of cardiac involvement, with no evidence of abnormal serum free light chains.
3. Have a diagnosis of cardiac amyloidosis within 2 years of screening. PART 3

   1. Understand the study procedures and agree to participate in the study by giving written informed consent as described in Section 10.1 - Appendix 1.
   2. Be male or female >18 years of age.
   3. WOCBP (those who have not been surgically sterilized, are not postmenopausal [i.e., last menstrual period > 2 years ago without pharmaceutical intervention], and women who are fertile) must have a negative pregnancy test prior within 24 h prior to infusion.
   4. WOCBP who are not exclusively in same-sex relationships and male participants with female sexual partners who are WOCBP must agree to use adequate contraceptive methods, defined as use of a condom by the male partner combined with use of a highly effective method of contraception by the female partner, for at least 2.5 days after injection of 99mTc-p5+14.
   5. Be in good general health, as determined by no clinically significant findings (including Type 2 diabetes mellitus) in the opinion of the Investigator from review of the medical history.
   6. Does not have a diagnosis of amyloidosis nor has a first- or second-degree relative (parent, sibling, child, aunt, uncle, niece, nephew) with confirmed or suspected familial amyloidosis.

PART 4

1. Understand the study procedures and agree to participate in the study by giving written informed consent as described in Section 10.1 - Appendix 1.
2. Be male or female >18 years of age.
3. Women of child-bearing potential (those who have not been surgically sterilized, are not postmenopausal [i.e., last menstrual period >2 years ago without pharmaceutical intervention], and women who are fertile) must have a negative pregnancy test prior within 24 h prior to infusion.
4. WOCBP who are not exclusively in same-sex relationships and male participants with female sexual partners who are WOCBP must agree to use adequate contraceptive methods, defined as use of a condom by the male partner combined with use of a highly effective method of contraception by the female partner, for at least 2.5 days after injection of 99mTc-p5+14..
5. Has a confirmed diagnosis of systemic ATTR amyloidosis, based on either a histologic confirmation of a cardiac biopsy containing deposits of apple-green birefringent, Congophilic material or extracardiac biopsy and imaging parameters (ECHO or CMR), or abnormal serum biomarkers indicative of cardiac involvement, with no evidence of abnormal serum free light chains.
6. Has a diagnosis of cardiac amyloidosis within 2 years of screening.
7. Has a negative 99mTc-PYP imaging study.

Exclusion Criteria:

PARTS 1-4

1. Due to annual dosimetry limitations, patients who have participated in another nuclear medicine amyloid imaging clinical trial protocol and received tracer injection in the last 6 months.
2. Is pregnant or breast-feeding.
3. Is mentally or legally incapacitated, has significant emotional problems at the time of the study, or has a history of psychosis.
4. Has a known allergy to potassium iodide.
5. Receiving hemodialysis or peritoneal dialysis.
6. Has severe claustrophobia or any medical condition that would prevent completion of the imaging protocol.
7. Has any illness that, in the opinion of the Investigator, might confound the results of the study or pose additional risk to the subject.
8. Has received heparin or heparin analogs (e.g., enoxaparin, dalteparin, fondaparinux) within seven (7) days prior to 99mTc-p5+14 administration.
9. Have previously received any dose of p5+14, in any form.
10. Have a QTc interval, using Bazett's formula (QTcB) of >480 ms, measured within six months prior to enrollment, or assessed prior to injection.
11. Have a serum AST >2x the upper limit of normal or 80 IU/L AND total bilirubin > 1.5x the upper limit of normal or 1.8 mg/dL within the previous six months of enrollment.
12. Have a serum ALT >2x the upper limit of normal or 64 IU/L AND total bilirubin > 1.5x the upper limit of normal or 1.8 mg/dL within the previous six months of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Whole body effective dosimetry measurement | From enrollment to the end of study is 8 days
  Whole body effective radiation dose assessed from analysis of organ-specific radioactivity uptake in planar and SPECT images.

SECONDARY OUTCOMES:
Measure cardiac uptake of 99mTc-p5+14 radioactivity from planar and SPECT/CT images in comparison to 99mTc-PYP uptake | From enrollment to the end of study is 8 days
  Measurement of 99mTc-p5+14 uptake in the heart of healthy volunteers and patients with systemic AL or ATTR amyloidosis and comparison with contemporaneous 99mTc-PYP cardiac radioactivity.
Measure uptake of 99mTc-p5+14 radioactivity in extracardiac tissues from planar and SPECT/CT images | From enrollment to the end of study is 8 days
  Measurement of 99mTc-p5+14 radioactivity in abdominothoracic organs of healthy volunteers and patients with systemic AL or ATTR amyloidosis from planar and SPECT/CT images.

OTHER OUTCOMES:
Compare planar and SPECT imaging of 99mTc-p5+14 for the detection of cardiac amyloid | From enrollment to the end of study is 8 days
  To compare the quantitative cardiac uptake of 99mTc-p5+14 and 99mTc-PyP in patients with systemic ATTR amyloidosis imaged by planar gamma scitigraphic and SPECT/CT imaging acquired at 1-hour and 3-hour post-injection.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Wall, PhD, Principal Investigator — University of Tennessee Graduate School of Medicine
Locations (1):
- University of Tennessee Graduate School of Medicine, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No